CLINICAL TRIAL: NCT00623194
Title: A 52-Week, Multinational, Multi-Centre, Open-Labelled Extension Trial of Insulin Detemir in Children and Adolescents 3-17 Years With Type 1 Diabetes on a Basal-Bolus Regimen With Insulin Aspart as Bolus Insulin
Brief Title: Safety Follow-up on Children and Adolescents With Type 1 Diabetes Treated With Insulin Detemir. An Extension to Trial NN304-1689
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN304-1690; 2006-002478-23 (EudraCT Number)
Record Dates: First submitted 2008-02-14; First posted 2008-02-25 (Estimated); Results first posted 2011-01-24 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Insulin Detemir; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- insulin detemir (Experimental): Insulin detemir up to twice daily plus insulin aspart at larger meals, doses are adjusted individually (treatment up to 104 weeks)
  Interventions: Drug: insulin detemir; Drug: insulin aspart

INTERVENTIONS:
Drug: insulin detemir — Treat-to-target dose titration scheme (individually adjusted), injection s.c. (under the skin), once or twice daily.
Drug: insulin aspart — Treat-to target dose titration scheme (individually adjusted), injection s.c. (under the skin), at larger meals.

SUMMARY:
This trial is conducted in Europe. The aim of this research is to assess the safety of continuous treatment with insulin detemir following participation in trial NN304-1689 (NCT00435019) on antibody development.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent obtained before any trial-related activities. (Trial-related activities are any procedure that would not have been performed during normal management of the subject). The parents or legal representative of the subject must sign and date the Informed Consent Form.
* Finalised 52 weeks of treatment with insulin detemir in trial NN304-1689.
* Fertile females (girls who have had their first menstrual period) must use adequate contraception (barrier methods, contraceptive pills or intrauterine device (IUD)) if there is any risk of pregnancy in the opinion of the Investigator. For Denmark and France only contraceptive pills or intrauterine device are considered as adequate contraceptive methods.

Exclusion Criteria:

* Significant concomitant disease such as endocrine, hepatic, renal, cardiac, respiratory, neurological, gastrointestinal, malignant or pancreatic diseases as judged by the Investigator.
* Pregnant or the intention of becoming pregnant.
* Previous participation in this trial (defined as enrolment).

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 146 (Actual)
Dates: Start 2008-02; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (30):
- Bulgaria (3):
  - Novo Nordisk Investigational Site, Pleven
  - Novo Nordisk Investigational Site, Sofia
  - Novo Nordisk Investigational Site, Varna
- Czechia (3):
  - Novo Nordisk Investigational Site, Olomouc
  - Novo Nordisk Investigational Site, Pardubice
  - Novo Nordisk Investigational Site, Prague
- Denmark (3):
  - Novo Nordisk Investigational Site, Glostrup Municipality
  - Novo Nordisk Investigational Site, Kolding
  - Novo Nordisk Investigational Site, Odense
- Finland (4):
  - Novo Nordisk Investigational Site, Helsinki
  - Novo Nordisk Investigational Site, Oulu
  - Novo Nordisk Investigational Site, Seinäjoki
  - Novo Nordisk Investigational Site, Turku
- France (2):
  - Novo Nordisk Investigational Site, Paris
  - Novo Nordisk Investigational Site, Toulouse
- Hungary (2):
  - Novo Nordisk Investigational Site, Budapest
  - Novo Nordisk Investigational Site, Miskolc
- Novo Nordisk Investigational Site, Skopje, North Macedonia
- Poland (3):
  - Novo Nordisk Investigational Site, Gdansk
  - Novo Nordisk Investigational Site, Kielce
  - Novo Nordisk Investigational Site, Warsaw
- Russia (2):
  - Novo Nordisk Investigational Site, Moscow
  - Novo Nordisk Investigational Site, Saint Petersburg
- Turkey (Türkiye) (4):
  - Novo Nordisk Investigational Site, Altunizade-Istanbul
  - Novo Nordisk Investigational Site, Antalya
  - Novo Nordisk Investigational Site, Istanbul
  - Novo Nordisk Investigational Site, Izmir
- United Kingdom (3):
  - Novo Nordisk Investigational Site, Aberdeen
  - Novo Nordisk Investigational Site, Dundee
  - Novo Nordisk Investigational Site, Norfolk

REFERENCES:
- [Background] Thalange N, Bereket A, Jensen LB, Hiort LC, Peterkova V. Development of Insulin Detemir/Insulin Aspart Cross-Reacting Antibodies Following Treatment with Insulin Detemir: 104-week Study in Children and Adolescents with Type 1 Diabetes Aged 2-16 Years. Diabetes Ther. 2016 Dec;7(4):713-724. doi: 10.1007/s13300-016-0196-5. Epub 2016 Sep 6. PMID 27600385
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 29 sites in 11 countries: (Bulgaria (3 sites), Czech Republic (3 sites), Denmark (2 sites), Finland (4 sites), France (1 site), Hungary (2 sites), Macedonia (1 site), Poland (4 sites), Russian Federation (4 sites), Turkey (4 sites) and United Kingdom (1 site)
Pre-assignment Details: At entry subjects had finalised 52-weeks treatment with insulin detemir plus insulin aspart (Trial NN304-1689, NCT00435019). Subjects treated with NPH insulin plus insulin aspart in trial NN304-1689 were not offered to continue in this extension trial. Subjects continued treatment with insulin detemir and insulin aspart doses from trial NN304-1689.
Period: Overall Study
Arm/Group | Insulin Detemir
Started | 146
Completed | 141
Not Completed | 5
Not completed — Lack of Efficacy | 1
Not completed — Protocol Violation | 3
Not completed — Unclassified | 1

BASELINE CHARACTERISTICS:
Arm/Group | Insulin Detemir
Number analyzed (Participants) | 146
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at entry in NN304-1689 (NCT00435019)
  years | 10.1 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77
  Male | 69
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 144
  More than one race | 0
  Unknown or Not Reported | 2
Age [Number; unit: participants] — Number of subjects in each age group at entry in NN304-1689 (NCT00435019)
  participants
    2-5 years | 37
    6-12 years | 59
    13-16 years | 50
Height [Mean (Standard Deviation); unit: meters] — Height at entry in NN304-1689 (NCT00435019)
  meters | 1.39 (0.26)
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index (BMI) at entry in NN304-1689 (NCT00435019)
  kg/m^2 | 18.14 (2.81)
Pubertal Status [Number; unit: participants] — Tanner scale:
  Pre-pubertal: Tanner grade 1: the vellus over the pubes is not further developed than that over the abdominal wall, i.e. no pubic hair.
  Pubertal: Tanner grade 2 or more: sparse growth of long slightly pigmented downy hair, straight, or slightly curled, chiefly at base of penis or along labia.
  participants
    Tanner grade 1 | 83
    Tanner grade 2+ | 63

OUTCOME MEASURES:

1. Primary Outcome: Insulin Detemir-insulin Aspart Cross-reacting Antibodies
Description: Estimated amount of bound antibodies in percent of total antibodies. The primary analysis of cross-reacting antibodies included results from blood samples taken before insulin detemir and less than 3 hours after insulin aspart injection. In addition, an analysis was done including results from samples taken before insulin detemir and less than 2.5 hours after insulin aspart injection.
Time Frame: week 0, 52 and 104
Population: Full analysis set 146 (100%), safety analysis set 146 (100%)
  The full analysis set was used for efficacy analyses and included subjects with signed informed consent who had been exposed to trial drug in extension.
  The safety analysis set included all subjects with a signed informed consent who were exposed in the extension.
Measure: Mean (Standard Error); unit: Percent bound of total
Arm/Group | Insulin Detemir
Number analyzed (Participants) | 146
Percent bound of total
  Week 0 (3 hours) | 31.11 (1.25)
  Week 52 (3 hours) | 43.99 (1.02)
  Week 104 (3 hours) | 35.96 (1.14)
  Week 0 (2.5 hours) | 31.22 (1.23)
  Week 52 (2.5 hours) | 44.09 (1.01)
  Week 104 (2.5 hours) | 35.92 (1.13)

2. Secondary Outcome: Development of Insulin Detemir Specific Antibodies and Insulin Aspart Specific Antibodies
Description: Amount of Insulin Detemir and Insulin Aspart specific antibodies in percent of total antibodies after 0, 52 and 104 weeks.
Time Frame: At 0, 52 and 104 weeks
Population: The safety analysis set included all subjects with a signed informed consent who were exposed in the extension period.
Measure: Mean (Standard Error); unit: Percent bound of total
Arm/Group | Insulin Detemir
Number analyzed (Participants) | 146
Percent bound of total
  Insulin Detemir specific, week 0 | 2.81 (1.28)
  Insulin Detemir specific, week 52 | 4.40 (1.27)
  Insulin Detemir specific, week 104 | 3.05 (1.27)
  Insulin Aspart specific, week 0 | 1.32 (0.67)
  Insulin Aspart specific, week 52 | 2.79 (0.64)
  Insulin Aspart specific, week 104 | 1.99 (0.65)

3. Secondary Outcome: Glycosylated Haemoglobin A1c (HbA1c)
Description: Glycosylated Haemoglobin A1c (HbA1c) measured after 104 weeks.
Time Frame: At 104 weeks
Population: Full analysis set 146 (100%) The full analysis set was used for efficacy analyses and included subjects with signed informed consent who had been exposed to trial drug in extension.
Measure: Mean (Standard Deviation); unit: Percent (%) glycosylated haemoglobin
Arm/Group | Insulin Detemir
Number analyzed (Participants) | 146
Percent (%) glycosylated haemoglobin | 8.74 (1.52)

4. Secondary Outcome: Fasting Plasma Glucose Values
Description: FPG (Fasting Plasma Glucose) values after 104 weeks.
Time Frame: At 104 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Insulin Detemir
Number analyzed (Participants) | 146
mmol/L | 7.71 (3.55)

5. Secondary Outcome: Hypoglycaemic Episodes
Description: Mild: signs/symptoms but able to treat him/herself. Moderate: signs/symptoms not able to treat him/herself. Responds to oral treatment.
  Severe: signs/symptoms and unable to treat him/herself. semiconscious/unconscious/in coma +/- convulsion and may require parenteral treatment.
Time Frame: Weeks 0-104
Population: The safety analysis set included all subjects with a signed informed consent who were exposed in the extension.
Measure: Number; unit: events
Arm/Group | Insulin Detemir
Number analyzed (Participants) | 146
events
  Overall, Mild | 10530
  Overall, Moderate | 450
  Overall, Severe | 7
  Overall, Biochemical | 5080
  Overall, Unclassified | 7
  Daytime, Mild | 9080
  Daytime, Moderate | 396
  Daytime, Severe | 3
  Daytime, Biochemical | 4122
  Daytime, Unclassified | 4
  Night-time, Mild | 1450
  Night-time, Moderate | 54
  Night-time, Severe | 4
  Night-time, Biochemical | 958
  Night-time, Unclassified | 3
  Total hypoglycaemic episodes | 16074
  Total hypoglycaemic episodes, daytime | 13605
  Total hypoglycaemic episodes, night-time | 2469

6. Secondary Outcome: BMI (Body Mass Index)
Description: BMI (Body Mass Index) after 104 weeks.
Time Frame: At 104 weeks
Population: The safety analysis set included all subjects with a signed informed consent who were exposed in the extension.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Insulin Detemir
Number analyzed (Participants) | 144
kg/m^2 | 18.88 (3.19)

7. Secondary Outcome: SD-score (Z-score) for Body Weight
Description: Standard deviation-score (SD-score) after 104 weeks. The SD-score for weight was calculated based on a British reference population from 1990. To estimate the growth of children, standardised mean weight values were calculated for each month of age and for each sex. Thus, a child with a weight equal to the mean value for its age and sex has an SD score of 0, while a child with a weight 2 SDs above the mean value for its age and sex has an SD score of +2.
Time Frame: At 104 weeks
Population: The safety analysis set included all subjects with a signed informed consent who were exposed in the extension.
Measure: Mean (Standard Deviation); unit: SD-scores
Arm/Group | Insulin Detemir
Number analyzed (Participants) | 144
SD-scores | 0.13 (0.97)

8. Secondary Outcome: Diabetic Ketoacidosis
Description: Diabetic ketoacidosis requiring hospitalisation
Time Frame: At 104 weeks
Population: The safety analysis set included all subjects with a signed informed consent who were exposed in the extension.
Measure: Number; unit: events
Arm/Group | Insulin Detemir
Number analyzed (Participants) | 146
events | 3

9. Secondary Outcome: Insulin Dose
Description: Daily insulin doses (basal (Insulin Detemir) and bolus (Insulin Aspart)) at week 104.
Time Frame: At 104 weeks
Population: The safety analysis set included all subjects with a signed informed consent who were exposed in the extension.
Measure: Mean (Standard Deviation); unit: U/kg
Arm/Group | Insulin Detemir
Number analyzed (Participants) | 144
U/kg
  Insulin Detemir dose (Basal) | 0.66 (0.29)
  Insulin Aspart dose (Bolus) | 0.51 (0.19)

10. Secondary Outcome: Laboratory Values: Albumin Serum and Total Protein Serum (g/dL)
Description: Albumin Serum and Total Protein Serum after 104 weeks.
Time Frame: At 104 weeks
Population: The safety analysis set included all subjects with a signed informed consent who were exposed in the extension.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Insulin Detemir
Number analyzed (Participants) | 144
g/dL
  Albumin serum (n=144) | 4.32 (0.25)
  Total Protein serum (n=144) | 7.09 (0.45)

11. Secondary Outcome: Laboratory Values: Creatine Serum Umol/L
Description: Creatine serum after 104 weeks.
Time Frame: At 104 weeks
Population: The safety analysis set included all subjects with a signed informed consent who were exposed in the extension.
Measure: Mean (Standard Deviation); unit: Umol/L
Arm/Group | Insulin Detemir
Number analyzed (Participants) | 144
Umol/L | 51.08 (13.55)

12. Secondary Outcome: Laboratory Values: Sodium Serum, Potassium Serum and Haemoglobin (mmol/L)
Description: Sodium Serum, Potassium Serum and Haemoglobin after 104 weeks.
Time Frame: At 104 weeks
Population: The safety analysis set included all subjects with a signed informed consent who were exposed in the extension.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Insulin Detemir
Number analyzed (Participants) | 144
mmol/L
  Sodium Serum (n=144) | 141.6 (3.11)
  Potassium serum (n=137) | 4.38 (0.50)
  Haemoglobin (n=144) | 8.28 (0.65)

13. Secondary Outcome: Laboratory Values: Alkaline Phosphatase Serum, Alanine Aminotransferase Serum and Lactate Dehydrogenase Serum (U/L)
Description: Alkaline phosphatase serum, Alanine Aminotransferase serum and Lactate Dehydrogenase serum after 104 weeks.
Time Frame: At 104 weeks
Population: The safety analysis set included all subjects with a signed informed consent who were exposed in the extension.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Insulin Detemir
Number analyzed (Participants) | 144
U/L
  Alkaline phosphatase serum (n=144) | 226.7 (197.10)
  Alanine Aminotransferase serum (n=144) | 19.0 (8.26)
  Lactate Dehydrogenase serum (n=137) | 199.6 (40.34)

14. Secondary Outcome: Laboratory Values: Leukocytes and Thrombocytes
Description: Leukocytes and Thrombocytes after 104 weeks.
Time Frame: At 104 weeks
Population: The safety analysis set included all subjects with a signed informed consent who were exposed in the extension.
Measure: Mean (Standard Deviation); unit: 10^9/L
Arm/Group | Insulin Detemir
Number analyzed (Participants) | 144
10^9/L
  Leukocytes (n=144) | 6.72 (1.85)
  Thrombocytes (n=144) | 301.90 (76.55)

15. Secondary Outcome: Fundoscopy/Fundus Photography
Description: Fundoscopy after 104 weeks. Abn. CS = Abnormal, clinically significant Abn. NCS = Abnormal, Not clinically significant
  Abn. CS = Abnormal, clinically significant Abn. NCS = Abnormal, Not clinically significant
Time Frame: at 52 weeks and at 104 weeks
Population: The safety analysis set included all subjects with a signed informed consent who were exposed in the extension.
Measure: Number; unit: participants
Arm/Group | Insulin Detemir
Number analyzed (Participants) | 146
participants
  Abnormal, clinically significant | 1
  Abnormal, not clinically significant | 8
  Normal | 131
  Missing | 6
  Abn CS baseline and 104 weeks | 1

16. Secondary Outcome: Vital Signs: Blood Pressure
Description: Blood pressure (Systolic and Diastolic) after 104 weeks.
Time Frame: At 104 weeks
Population: The safety analysis set included all subjects with a signed informed consent who were exposed in the extension.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Insulin Detemir
Number analyzed (Participants) | 143
mmHg
  Systolic Blood Pressure | 109.5 (13.6)
  Diastolic Blood Pressure | 66.6 (8.9)

17. Secondary Outcome: Vital Signs: Pulse
Description: Pulse at week 104
Time Frame: At 104 weeks
Population: The safety analysis set included all subjects with a signed informed consent who were exposed in the extension.
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | Insulin Detemir
Number analyzed (Participants) | 141
beats/minute | 82.6 (9.0)

ADVERSE EVENTS:
Time Frame: The adverse events were collected over a period of 104 weeks.
Description: The safety analysis set is all subjects exposed to at least one dose of trial drug.
Arm/Group | Insulin Detemir
Serious Adverse Events (participants affected / at risk) | 12/146
Other Adverse Events (participants affected / at risk) | 108/146
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Detemir (N=146)
Gastroenteritis (Infections and infestations) | 2 (2)
Abscess limb (Infections and infestations) | 1 (1)
Gastroenteritis shigella (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Otitis media acute (Infections and infestations) | 1 (1)
Soft tissue infection (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 3 (3)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (3)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1)
Hypoglycaemia unconsciousness (Metabolism and nutrition disorders) | 1 (1)
Burns second degrees (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Detemir (N=146)
Nasopharyngitis (Infections and infestations) | 71 (164)
Upper Respiratory Tract Infection (Infections and infestations) | 21 (44)
Pharyngitis (Infections and infestations) | 20 (41)
Influenza (Infections and infestations) | 17 (38)
Gastroenteritis (Infections and infestations) | 15 (21)
Bronchitis (Infections and infestations) | 9 (16)
Viral infection (Infections and infestations) | 10 (12)
Rhinitis (Infections and infestations) | 9 (11)
Acute Tonsilliitis (Infections and infestations) | 8 (8)
Headache (Nervous system disorders) | 25 (84)
Abdominal pain upper (Gastrointestinal disorders) | 8 (13)
Abdominal pain (Gastrointestinal disorders) | 9 (10)
Vomiting (Gastrointestinal disorders) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk reserves the right not to release data until specified milestones, e.g., a Clinical Trial Report is available. At the end of the trial, one or more manuscripts for publication will be prepared in collaboration between authors and Novo Nordisk. Novo Nordisk will not suppress or veto publications; however Novo Nordisk reserves the right to postpone publication and/or communication for a short time to protect intellectual property.